CLINICAL TRIAL: NCT03590925
Title: Evaluation of the Improvement of Primary Prevention in Ischemic Cardiomyopathy Patients Using New Screening and Referring System (Advance-ICM)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0075
Record Dates: First submitted 2018-06-19; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- new screening and referring system of ICD: Non-randomized, non-blinded, multi-center study receiving new screening and referring system of ICD

SUMMARY:
The patients who undergo ICD(implantable cardioverter defibrillator) implantation for the primary prevention of sudden cardiac death with severe LV(left ventricle) dysfunction (ejection fraction ≤ 40%) by ICM(idiopathic cardiomyopathy).

Indications for ICD implantation for primary prevention in accordance with 2016 revised Korean indication guideline on ICD implantation

* FU LVEF(Left Ventricular Ejection Fraction) ≤ 30% (at least 40 days post-myocardial infarction)
* FU LVEF 31~35%, NYHA(the New York Heart Association) class II, III (at least 40 days post-myocardial infarction)
* FU LVEF ≤ 40%, NSVT(non-sustained ventricular tachycardia) (Holter), inducible VF(ventricular flutter) or sustained VT(ventricular tachycardia) at electrophysiological study (at least 40 days post-myocardial infarction)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Patients eligible for the indications for ICD implantation for primary prevention indication in accordance with 2016 revised Korean indication guideline on ICD implantation
* Patients should be managed by non-EP physician
* Patients who are willing to sign the informed consent
* Patients who are willing to receive the implantation and post-operative follow-up

Exclusion Criteria:

* Malignant tumor
* Life expectancy < 12 months
* Patients unable or unwilling to cooperate in the study procedures

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who undergo ICD implantation for the primary prevention of sudden cardiac death with severe LV dysfunction (ejection fraction ≤ 40%) by ICM.
  Indications for ICD implantation for primary prevention in accordance with 2016 revised Korean indication guideline on ICD implantation
  * FU LVEF ≤ 30% (at least 40 days post-myocardial infarction)
  * FU LVEF 31~35%, NYHA class II, III (at least 40 days post-myocardial infarction)
  * FU LVEF ≤ 40%, NSVT (Holter), inducible VF or sustained VT at electrophysiological study (at least 40 days post-myocardial infarction)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of the quality of care in patients with ICM | 3 years
  the rate of device therapy(ICD or CRT-D(Cardiac Resynchronization Therapy-Device))

SECONDARY OUTCOMES:
Improvement of the cardiovascular outcome of patients | 3 years
  Cardiovascular outcome (cardiovascular death, Non-cardiovascular death)
Improvement of the cardiovascular outcome of patients | 3 years
  Pattern of arrhythmia measured by EKG or echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Yu HT, Oh IY, Choi EK, Sung JH, Lee YS, Kim JY, Baek Y, Park J, Joung B; ADVANCE-ICM investigators. Clinical and Hospital Factors Affecting Treatment with Primary Prevention Implantable Cardioverter-Defibrillators in Ischemic Cardiomyopathy Patients. Yonsei Med J. 2020 Nov;61(11):942-950. doi: 10.3349/ymj.2020.61.11.942. PMID 33107237